CLINICAL TRIAL: NCT06950723
Title: Efficacy of Chest Physical Therapy on Arterial Blood Gases for Neonates Post Hypoxic Ischemic Encephalopathy in Neonatal Intensive Care Unit: A Clinical Trial Study
Brief Title: Chest Physical Therapy on Arterial Blood Gases for Neonates Post Hypoxic Ischemic Encephalopathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Elsayed Mehrem, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Sayed75
Record Dates: First submitted 2025-04-09; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Hypoxic Ischemic Encephalopathy of Newborn
MeSH Terms: interventions — 2-cyclohexylidenhydrazo-4-phenyl-thiazole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chest physical Therapy group (Experimental): Study group
  Interventions: Other: Chest Physical Therapy (CPT) modalities , Medical Treatment
- Medical treatment group (Experimental): Control group
  Interventions: Other: Chest Physical Therapy (CPT) modalities , Medical Treatment

INTERVENTIONS:
Other: Chest Physical Therapy (CPT) modalities , Medical Treatment — Chest Physical Therapy (CPT) modalities in the form of postural drainage, percussion and vibration.

SUMMARY:
Hypoxic-ischemic encephalopathy (HIE) is a dangerous illness that happens when a newborn's brain does not receive adequate oxygen and blood flow, which can result in serious effects such as cerebral palsy and epilepsy. Infant diagnosed with HIE required ventilator support and subsequently developed pneumonia. They experienced respiratory problems and feeding challenges. Chest Physical Therapy is the best modalities to clear chest and improve ventilation.

DETAILED DESCRIPTION:
The purpose of this study to investigate the effect of chest physical therapy on Arterial Blood Gases for neonates post hypoxic ischemic encephalopathy (HIE) in Neonatal intensive care unit.

Methods: Fifty neonates from both sexes, age from birth to 10 days, post HIE with chest problems were selected from neonatal intensive care unit (NICU) at Minia University hospital, Egypt. They were divided into two equal groups, control group (CG) received traditional medical treatment according to American Academy of Pediatrics (AAP) recommendations and study group (SG) received traditional medical treatment plus Chest Physical Therapy (CPT) modalities in the form of postural drainage, percussion and vibration. The sessions will apply once daily for 6 days/week, each session is about 30 minutes, according to the neonate tolerance till complete clinical cure and discharge from NICU.

the outcome will measure by Timing of Arterial blood gases improvement, Duration required for clinical improvement, Duration of Mechanical ventilation, Duration of Hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Neonates with chest problems post Hypoxic-ischemic encephalopathy

Exclusion Criteria:

* Neonates with chest problems due to other Causes except post Hypoxic-ischemic encephalopathy.
* unstable medical status
* Neonates with Post-operative s' respiratory problems due to any reasons.

Ages: 1 Day to 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-05-10 (Estimated); Primary Completion 2025-06-10 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Timing of Arterial blood gases improvement | 3-14 days
  Time needed to improve Arterial blood gases due to CPT
Timing required for clinical improvement | 3-14 days
  Time needed to improve clinical signs due to CPT
Timing needed for Mechanical Ventilation | 3-7 days
  Time needed to Mechanical Ventilation support.
Hospitalization time | 5-21 days
  All staying duration need for the neonates from admission till discharge from the hospital.